CLINICAL TRIAL: NCT03982368
Title: A 4 Weeks, Phase II, Multicenter, Randomized, Double-masked, Vehicle-controlled, Parallel Group Study With 12 Weeks of Follow-up to Evaluate Safety and Efficacy of rhNGF Eye Drops Solution vs Vehicle in Moderate to Severe Dry Eye.
Brief Title: A Study to Evaluate Safety and Efficacy of rhNGF Eye Solution vs Vehicle in Patients With Moderate to Severe Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGF0118
Record Dates: First submitted 2019-05-23; First posted 2019-06-11 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — cenegermin

STUDY DESIGN:
Intervention Model Description: Parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- rhNGF 20 μg/ml TID (Experimental): One drop of rhNGF 20 μg/ml will be instilled in both eyes three times daily (every 6-8 hours)
  Interventions: Drug: rhNGF 20 μg/ml
- rhNGF 20 μg/ml BID + vehicle OD (Experimental): One drop of rhNGF 20 μg/ml will be instilled in both eyes two times daily (BID) plus one drop (40 μL) of vehicle will be instilled in both eyes once daily (OD) (every 6-8 hours)
  Interventions: Drug: rhNGF 20 μg/ml + vehicle
- Vehicle TID (Placebo Comparator): Vehicle eye one drop will be instilled in both eyes three times daily (every 6-8 hours)
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: rhNGF 20 μg/ml — one drop of rhNGF 20 μg/ml will be instilled in both eyes three times daily (every 6-8 hours)
  Other Names: cenegermin
  Arms: rhNGF 20 μg/ml TID
Drug: rhNGF 20 μg/ml + vehicle — one drop of rhNGF 20 μg/ml will be instilled in both eyes two times daily plus one drop (40 μL) of vehicle will be instilled in both eyes once daily (every 6-8 hours).
  rhNGF will be instilled in the morning and in the evening while the vehicle will be instilled in the afternoon.
  Other Names: cenegermin + placebo
  Arms: rhNGF 20 μg/ml BID + vehicle OD
Other: Vehicle — one drop of vehicle will be instilled in both eyes three times daily (every 6-8 hours)
  Other Names: placebo
  Arms: Vehicle TID

SUMMARY:
The objective of this study is to assess the efficacy and safety of rhNGF eye drops at 20 μg/ml concentration administered two or three times daily for 4 weeks in patients with moderate to severe dry eye.

DETAILED DESCRIPTION:
This is a 4 weeks, Phase II, multicenter, randomized, double-masked, vehicle-controlled, parallel group study with 12 weeks of follow-up, designed to perform dose-ranging and to evaluate safety and efficacy of recombinant human Nerve Growth Factor (rhNGF) eye drops solution versus vehicle, in patients with moderate to severe dry eye (DE).

Test product is rhNGF 20 μg/ml; reference product is vehicle. Test and reference will be instilled in both eyes according to the following scheme:

Group 1: one drop of rhNGF 20 μg/ml is instilled in both eyes three times daily (every 6-8 hours, e.g. 7:00 am, 02:00 pm; 09:00 pm).

Group 2: one drop of rhNGF 20 μg/ml is instilled in both eyes two times daily (in the morning and in the evening) plus one drop (40 μL) of vehicle (placebo) is instilled in both eyes once daily in the afternoon.

Group 3: one drop (40 μL) of vehicle (placebo) is instilled in both eyes three times daily (every 6-8 hours, e.g. 7:00 am, 02:00 pm; 09:00 pm).

Approximate randomization 1:1:1 of 261 patients to rhNGF eye drops solution 20 μg/ml TID (87 patients) or rhNGF eye drops solution 20 μg/ml BID + vehicle eye drop SID (86 patients) or vehicle eye drops solution (88 patients) TID for 4 weeks was applied.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years
2. Patients with moderate to severe dry eye characterized by the following clinical features:

   1. Corneal and/or conjunctival staining with fluorescein using National Eye Institute (NEI) grading system > 3
   2. SANDE questionnaire >25 mm
   3. Schirmer test I (without anaesthesia) >2mm <10 mm/5 minutes
   4. Tear film break-up time (TFBUT) < 10 seconds in the worse eye
3. The same eye (eligible eye) must fulfill all the above criteria
4. Patients diagnosed with dry eye at least 6 months before enrolment (current use or recommended use of artificial tears for the treatment of Dry Eye)
5. Best corrected distance visual acuity (BCDVA) score of ≥ 0.1 decimal units (20/200 Snellen value) in both eyes at the time of study enrolment
6. If a female of childbearing potential, have a negative pregnancy test
7. Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or legal representative must have been approved by the Institutional Review Board (IRB) / Independent Ethics Committee (IEC) for the current study
8. Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

1. Inability to speak and understand the local language sufficiently to understand the nature of the study, to provide written informed consent, and to allow the completion of all study assessments;
2. Evidence of an active ocular infection, in either eye
3. Presence of any other ocular disorder or condition requiring topical medication during the entire duration of study
4. History of severe systemic allergy or of ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis and/or keratitis other than dry eye
5. Intraocular inflammation defined as Tyndall score >0
6. History of malignancy in the last 5 years
7. Systemic disease not stabilized within 1 month before Screening Visit (e.g. diabetes with glycemia out of range, thyroid malfunction..) or judged by the investigator to be incompatible with the study (e.g. current systemic infections) or with a condition incompatible with the frequent assessment required by the study
8. Patient had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds or had a clinically significant allergy to drugs, foods, amide local anaesthetics or other materials including commercial artificial tears (in the opinion of the investigator)
9. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

   1. are currently pregnant or,
   2. have a positive result at the urine pregnancy test (Baseline/Day 0) or,
   3. intend to become pregnant during the study treatment period or,
   4. are breast-feeding or,
   5. are not willing to use highly effective birth control measures, such as: hormonal contraceptives - oral, implanted, transdermal, or injected - and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or Intra Uterine Device (IUD) - during the entire course of and 30 days after the study treatment periods
10. Any concurrent medical condition, that in the judgment of the PI, might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being
11. Use of topical cyclosporine, topical corticosteroids or any other topical drug for the treatment of dry eye in either eye within 30 days of study enrolment.
12. Contact lenses or punctum plug use during the study (previous use not an exclusion criteria but must be discontinued at the screening visit)
13. History of drug addiction or alcohol abuse
14. Any prior ocular surgery (including refractive palpebral and cataract surgery) if within 90 days before the screening visit
15. Participation in a clinical trial with a new active substance during the past 6 months
16. Participation in another clinical trial study at the same time as the present study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, PhD, Study Director — Dompé Farmaceutici SpA; William Lipsky, MD, Principal Investigator — Advanced Laser Vision Surgical Institute (Study Site) Intouch Clinical Research Center (SMO)
Locations (12):
- United States (12):
  - Global Research Management, Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Sierra Clinical Trials & Research Organization, Santa Ana, California
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Kentucky Eye Institute, Lexington, Kentucky
  - Tauber Eye Center, Kansas City, Missouri
  - Moyes Eye Center, Kansas City, Missouri
  - SightMD, Babylon, New York
  - Toyos Clinic, Nashville, Tennessee
  - Houston Eye Associates HEA - Gramercy Location, Houston, Texas
  - Advanced Laser Vision Surgical Institute (Study Site) Intouch Clinical Research Center (SMO), Houston, Texas

REFERENCES:
- [Derived] Wirta D, Lipsky W, Toyos M, Martel J, Goosey J, Verachtert A, El-Harazi S, Karpecki P, Allegretti M, Goisis G, Pasedis G, Mantelli F. Recombinant human nerve growth factor (cenegermin) for moderate-to-severe dry eye: phase II, randomized, vehicle-controlled, dose-ranging trial. BMC Ophthalmol. 2024 Jul 17;24(1):290. doi: 10.1186/s12886-024-03564-w. PMID 39020305

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment of a total of 300 patients was planned. Due to restrictions in the hospital clinical routines related to coronavirus disease 2019, the sponsor decided to prematurely stop enrollment in the study in order to comply with quarantine measures of each country and avoid risks of infection of COVID-19 illness for all involved patients.
  A total of 261 patients were randomized to receive study treatment: 87 in the rhNGF TID group, 86 in the rhNGF BID group, and 88 in the vehicle TID group.
Groups:
- rhNGF 20 μg/ml BID + Vehicle OD: One drop of rhNGF 20 μg/ml will be instilled in both eyes two times daily (BID) plus one drop (40 μL) of vehicle will be instilled in both eyes once daily (OD) (every 6-8 hours)
  rhNGF 20 μg/ml + vehicle: one drop of rhNGF 20 μg/ml will be instilled in both eyes two times daily plus one drop (40 μL) of vehicle will be instilled in both eyes once daily (every 6-8 hours).
  rhNGF will be instilled in the morning and in the evening while the vehicle will be instilled in the afternoon.
Period: Overall Study
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Started | 87 | 86 | 88
FAS Popuation (The FAS consisted of all patients randomized who took at least 1 dose of IMP and who had at least 1 postbaseline efficacy measurement for the primary endpoint. This analysis set was used for the primary efficacy analysis. Patients were analyzed according to the randomized treatment.) | 81 | 82 | 84
PP Population (The PP set consisted of all patients in the FAS who fulfilled the study protocol requirements in terms of IMP intake and collection of primary efficacy data and had no major deviations that may have affected study results. This analysis set was used for supportive efficacy analysis.) | 72 | 71 | 80
Completed | 74 | 79 | 83
Not Completed | 13 | 7 | 5
Not completed — Adverse Event | 6 | 4 | 3
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — unknow | 4 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): The FAS consisted of all patients randomized who took at least 1 dose of IMP and who had at least 1 postbaseline efficacy measurement for the primary endpoint.
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID | Total
Number analyzed (Participants) | 81 | 82 | 84 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 54 | 61 | 166
  >=65 years | 30 | 28 | 23 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (13.52) | 60.2 (12.39) | 59.1 (11.50) | 60.4 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 69 | 72 | 198
  Male | 24 | 13 | 12 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 13 | 37
  Not Hispanic or Latino | 66 | 73 | 71 | 210
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 81 | 82 | 84 | 247

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schirmer I Test (Without Anesthesia) vs Week 4 - Full Analysis Set
Description: The Schirmer test is used in ophthalmic examination to measure tear production for the diagnosis of conditions such as keratoconjunctivitis sicca and dry eye.
  Without previously instilling anesthetic drops, the Schirmer strip is inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters is recorded after 5 minutes.
  The patients will be instructed to close their eyes gently. After 5 minutes have elapsed, the Schirmer test strip will be removed and the length of the tear absorption on the strip will be measured (millimeters/5 minutes)
  Cutoff values:
  <5 mm - pathologic dry eye 5-10 mm - marginal dry eye >10 and <30 mm - normal secretion
Time Frame: Baseline, week 4
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
mm | 2.60 (0.77) | 3.99 (0.76) | 1.68 (0.75)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; The primary endpoint was analyzed using analysis of variance (ANOVA) including only treatment as the main factor, followed by preplanned comparisons from vehicle and rhNGF dosages according to Williams' procedure; Test type: Superiority; p = 0.078, ANOVA; least square mean difference = 0.93, 95% CI 2-sided [-1.47 to 3.32]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.066, ANOVA; least square mean difference = 2.31, 95% CI 2-sided [-0.08 to 4.70]

2. Primary Outcome: Change From Baseline in Schirmer I Test (Without Anesthesia) vs Week 4 - Per Protocol Set
Description: as for outcome 1
Time Frame: Baseline, week 4
Population: Per protocol (PP) set: The PP set consisted of all patients in the FAS who fulfilled the study protocol requirements in terms of IMP intake and collection of primary efficacy data and had no major deviations that may have affected study results.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
mm | 2.99 (0.78) | 3.72 (0.79) | 1.28 (0.74)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.032, ANOVA; Least square mean difference = 1.71, 95% CI 2-sided [-0.70 to 4.12]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.029, ANOVA; Least square mean difference = 2.44, 95% CI 2-sided [0.02 to 4.86]

3. Secondary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Scores for Severity vs Week 4 - Full Analysis Set
Description: The SANDE (symptom assessment in dry eye) score is composed by two questions presented in visual analog scale. The two questions assess the frequency and severity of dry eye syndrome. The global score is calculated by taking the square root of the product of the severity of symptoms per the frequency of symptoms. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
Time Frame: Baseline, week 4
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
score on a scale | -24.6 (27.15) | -20.3 (24.91) | -22.2 (22.29)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.534, t-test, 2 sided
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.611, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Scores for Severity vs Week 4 - Per Protocol Set
Description: as for outcome 3
Time Frame: Baseline, week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
score on a scale | -24.9 (27.35) | -19.9 (25.34) | -22.1 (21.74)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.486, t-test, 2 sided
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.564, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Scores for Frequency vs Week 4 - Full Analysis Set
Description: The SANDE (symptom assessment in dry eye) score is composed by two questions presented in visual analog scale. The two questions assess the frequency and severity of dry eye syndrome.The SANDE global score is calculated by taking the square root of the product of the frequency of symptoms and the severity of symptoms. The SANDE scale ranges from 0 to 100 wi.100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms
Time Frame: Baseline, week 4
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
score on a scale | -24.9 (26.29) | -22.7 (25.42) | -24.0 (23.81)

6. Secondary Outcome: Change From Baseline in Symptoms Questionnaire (SANDE) Scores for Frequency vs Week 4 - Per Protocol Set
Description: The SANDE (symptom assessment in dry eye) score is composed by two questions presented in visual analog scale. The two questions assess the frequency and severity of dry eye syndrome. The SANDE score is calculated by taking the square root of the product of the frequency of symptoms score. The SANDE scale ranges from 0 to 100 wi.100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
Time Frame: Baseline, week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
score on a scale | -24.7 (26.73) | -22.2 (25.67) | -23.8 (23.92)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.810, t-test, 2 sided
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.733, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Schirmer II Test (With Anesthesia) vs Week 4 - Full Analysis Set
Description: The Schirmer II test is performed as the Schirmer I test after instilling anesthetic drops. The Schirmer strips are inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters is recorded after 5 minutes. All patients are seated at rest with their eyes closed, and the lower cul-de-sac is gently dried with a cotton applicator before the placement of strips.
  Cut-off values:
  <5 mm - pathologic dry eye 5-10 mm - marginal dry eye >10 and <30 mm - normal secretion
Time Frame: Baseline, week 4
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
mm | 2.19 (0.69) | 0.89 (0.69) | 0.21 (0.68)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; The secondary endpoint was analyzed using analysis of variance (ANOVA) including only treatment as the main factor, followed by preplanned comparisons from vehicle and rhNGF dosages according to Williams' procedure; Test type: Superiority; p = 0.025, ANOVA; Least square mean difference = 1.97, 95% CI 2-sided [-0.19 to 4.13]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.243, ANOVA; Least square mean difference = 0.68, 95% CI 2-sided [-1.48 to 2.83]

8. Secondary Outcome: Change From Baseline in Schirmer II Test (With Anesthesia) vs Week 4 - Per Protocol Set
Description: as for outcome 7
Time Frame: Baseline, week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
mm | 2.24 (0.69) | 0.54 (0.70) | -0.18 (0.66)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.007, ANOVA; Least square mean difference = 2.41, 95% CI 2-sided [0.28 to 4.54]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.230, ANOVA; Least square mean difference = 0.71, 95% CI 2-sided [-1.43 to 2.85]

9. Secondary Outcome: Change From Baseline in Corneal and Conjunctiva Vital Staining With Fluorescein (National Eye Institute [NEI] Scales) vs Week 4 - Full Analysis Set
Description: Corneal staining total score is defined as the sum of scores from 5 corneal areas: Central, Superior, Temporal, Nasal, and Inferior. The score for each area ranges from 0 to 3 where grade 0 reflects normal/healthy situation, whereas grade 3 reflects a severe damage. Thus, the corneal staining total score can range from 0 to 15 where the higher the score the worse is the outcome.
  The conjunctiva is divided into a superior paralimbal area, an inferior paralimbal area and a peripheral area with a grading scale of 0-3 where grade 0 reflects normal/healthy situation, whereas grade 3 reflects a severe damage and with a maximal score of 9 for the nasal and temporal conjunctiva. Thus, the conjunctival staining total score can range from 0 to 18 where the higher the score the worse is the outcome.
  Corneal and conjunctiva vital staining total score is the sum of corneal staining total score and conjunctiva total score.
Time Frame: Baseline, week 4
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
score on a scale
  corneal and conjunctival total score | -3.75 (0.63) | -2.95 (0.62) | -2.60 (0.61)
  corneal score: number analyzed (Participants) | 78 | 81 | 84
  corneal score | -1.9 (2.84) | -1.8 (2.72) | -1.5 (2.92)
  conjunctiva score: number analyzed (Participants) | 76 | 79 | 82
  conjunctiva score | -2.1 (3.17) | -1.2 (3.58) | -1.4 (3.36)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; The secondary endpoint was analyzed using analysis of variance (ANOVA) including only treatment as the main factor, followed by preplanned comparisons from vehicle and rhNGF dosages according to Williams' procedure. p value for total corneal ancd conjunctival score is reported; Test type: Superiority; p = 0.799, ANOVA; Last Observation Carried Forward (LOCF) was used for imputing missing data in the Full analysis set at Week 4; Least square mean difference = -1.16, 95% CI 2-sided [-3.11 to 0.80]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.715, ANOVA; Least square mean difference = -0.36, 95% CI 2-sided [-2.30 to 1.59]

10. Secondary Outcome: Change From Baseline in Corneal and Conjunctiva Vital Staining With Fluorescein (National Eye Institute [NEI] Scales) vs Week 4 - Per Protocol Set
Description: as for outcome 9
Time Frame: Baseline, week 4
Population: Per protocol (PP) set: The PP set consisted of all patients in the FAS who fulfilled the study protocol requirements in terms of IMP intake and collection of primary efficacy data and had no major deviations that may have affected study results. This analysis set was used for supportive efficacy analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
score on a scale
  Total score | -3.94 (0.60) | -2.61 (0.61) | -2.40 (0.57)
  Corneal score | -1.9 (2.80) | -1.8 (2.61) | -1.5 (2.85)
  Conjunctival score | -1.9 (2.95) | -1.0 (3.05) | -1.3 (3.32)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.831, ANOVA; Least square mean difference = -1.54, 95% CI 2-sided [-3.40 to 0.31]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.750, ANOVA; Least square mean difference = -0.21, 95% CI 2-sided [-2.07 to 1.66]

11. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) vs Week 4 - Full Analysis Set
Description: Tear film break-up time (TFBUT) is the time taken to appear first dry spot on cornea after a complete blinking. TFBUT measurement is an easy and fast method used to assess the stability of tear film. It is a standard diagnostic procedure in the dry eye clinics. TFBUT is measured by determining the time to tear break-up. The TFBUT is performed after instillation of 5 μL of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. The patient is instructed to blink several times to thoroughly mix the fluorescein with the tear film.
  A TFBUT greater than 15 seconds is considered normal, while a break time of less than 10 seconds is to be considered pathological.
Time Frame: Baseline, week 4
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
seconds | 1.11 (0.25) | 0.43 (0.25) | 0.15 (0.25)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.004, ANOVA; Least square mean difference = 0.96, 95% CI 2-sided [0.17 to 1.75]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.217, ANOVA; Least square mean difference = 0.28, 95% CI 2-sided [-0.51 to 1.07]

12. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT) vs Week 4 - Per Protocol Set
Description: as for outcome 11
Time Frame: Baseline, week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
seconds | 1.11 (0.27) | 0.47 (0.27) | 0.19 (0.25)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.007, ANOVA; Least square mean difference = 0.92, 95% CI 2-sided [0.10 to 1.74]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.225, ANOVA; Least square mean difference = 0.28, 95% CI 2-sided [-0.54 to 1.10]

13. Secondary Outcome: Number of Patients Who Experienced a Worsening in Symptom Scores (SANDE) and/or NEI Score ≥ 50% Assessed at Week 4 - Full Analysis Set
Description: The SANDE score is calculated by taking the square root of the product of the severity of symptoms score. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms.
  The NEI/Industry Workshop guidelines are used for grading the scale of corneal and conjunctival damage.
  The cornea is divided into five sectors (central, superior, inferior, nasal and temporal), each of which is scored on a scale of 0-3, with a maximal total corneal staining score of 15.
  Both nasally and temporally, the conjunctiva is divided into a superior paralimbal area, an inferior paralimbal area, and a peripheral area with a grading scale of 0-3 and with a maximal total score of 9 for the nasal and temporal conjunctiva (overall the total score ranged from 0-18).
  Briefly, grade 0 reflects normal/healthy situation, whereas grade 3 reflects a severe damage in the considered sector.
Time Frame: At week 4
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
Participants | 2 | 9 | 3
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.680, t-test, 2 sided
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.066, t-test, 2 sided

14. Secondary Outcome: Number of Patients Who Experienced a Worsening in Symptom Scores (SANDE) and/or NEI Score ≥ 50% Assessed at Week 4 - Per Protocol Set
Description: as for outcome 13
Time Frame: At week 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
Participants | 0 | 8 | 3
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.097, Chi-squared
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.076, Chi-squared

15. Secondary Outcome: Change From Baseline in Quality of Life (Impact of Dry Eye on Everyday Life (IDEEL) Questionnaire vs Different Timepoints - Full Analysis Set
Description: IDEEL assesses quality of life, symptoms and treatment effects on patients with dry eye.
  The IDEEL contains 3 modules (Daily Activities, Treatment Satisfaction, and Symptom Bother) with a total of 57 questions.
  1. The Daily Activities Module is the quality of life instrument. It is comprised of 27 items.
  2. The IDEEL Treatment Satisfaction and Bother Module is divided into 2 sections, Treatment - In General and Treatment - Eye Drops.
  3. The Symptom Bother Module consists of 20 items in a single content domain, Symptom Bother.
  Scores for each dimensions ranged from 0 to 100.
  Higher scores for:
  * dimension of the Dry Eye Impact on Daily Life module indicates less impact on daily activities;
  * symptom-bother dimension indicates greater bother due to symptoms;
  * satisfaction with Treatment Effectiveness dimension indicates greater satisfaction with treatment effectiveness;
  * treatment-related bother/inconvenience indicates less treatment-related bother or inconvenience.
Time Frame: At weeks 4, 8, 12 and 16
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
score on a scale
  Daily activity limitations - Chance from baseline to week 4 | 16.5 (20.71) | 19.5 (17.55) | 13.1 (20.60)
  Daily activity limitations - Chance from baseline to week 8 | 16.8 (23.49) | 14.8 (18.07) | 11.2 (17.54)
  Daily activity limitations - Chance from baseline to week 12 | 15.7 (21.10) | 15.5 (20.01) | 11.1 (17.45)
  Daily activity limitations - Chance from baseline to week 16 | 14.2 (20.05) | 14.4 (21.23) | 9.4 (16.74)
  Emotional well-being - change from baseline to week 4 | 14.5 (21.18) | 16.3 (20.40) | 15.0 (20.47)
  Emotional well-being - change from baseline to week 8 | 16.2 (21.33) | 13.4 (18.64) | 12.7 (17.69)
  Emotional well-being - change from baseline to week 12 | 14.2 (18.66) | 15.3 (17.95) | 14.2 (18.20)
  Emotional well-being - change from baseline to week 16 | 16.0 (18.54) | 15.5 (19.17) | 13.5 (20.22)
  work limitations - change from baseline to week 4 | 16.3 (27.13) | 20.6 (24.29) | 17.4 (24.09)
  work limitations - change from baseline to week 8 | 18.0 (24.94) | 18.3 (19.00) | 17.0 (22.52)
  work limitations - change from baseline to week 12 | 16.4 (22.39) | 20.9 (22.05) | 17.8 (22.35)
  work limitations - change from baseline to week 16 | 16.3 (20.75) | 20.9 (20.83) | 16.0 (21.63)
  Treatment satisfaction/happiness - change from baseline to week 4 | 24.1 (30.81) | 19.0 (30.57) | 24.1 (33.57)
  Treatment satisfaction/happiness - change from baseline to week 8 | 28.8 (28.56) | 19.1 (26.90) | 13.3 (30.69)
  Treatment satisfaction/happiness - change from baseline to week 12 | 26.1 (30.30) | 19.1 (27.86) | 15.0 (26.83)
  Treatment satisfaction/happiness - change from baseline to week 16 | 26.1 (26.62) | 23.5 (29.29) | 12.7 (27.03)
  treatment-related bother - change from baseline to week 4 | 14.6 (22.78) | 16.8 (25.00) | 13.8 (27.19)
  treatment-related bother - change from baseline to week 8 | 10.6 (20.61) | 6.5 (26.56) | 4.8 (26.59)
  treatment-related bother - change from baseline to week 12 | 10.3 (22.71) | 8.7 (24.91) | 9.0 (27.95)
  treatment-related bother - change from baseline to week 16 | 10.8 (20.65) | 8.1 (23.88) | 10.0 (27.14)
  Dry eye symptom bother - change from baseline to week 4 | -16.8 (17.80) | -17.7 (16.54) | -16.5 (17.04)
  Dry eye symptom bother - change from baseline to week 8 | -21.2 (19.56) | -16.6 (15.46) | -13.5 (15.01)
  Dry eye symptom bother - change from baseline to week 12 | -19.6 (17.41) | -18.2 (17.30) | -13.0 (13.01)
  Dry eye symptom bother - change from baseline to week 16 | -19.9 (15.62) | -19.1 (17.75) | -11.1 (14.46)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Daily Activity Limitations - change from baseline to week 4; Test type: Superiority; p = 0.289, ANOVA; Least square mean difference = 16.4, 95% CI 2-sided [12.0 to 20.8]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 4; Test type: Superiority; p = 0.032, ANOVA; Least square mean difference = 19.7, 95% CI 2-sided [15.4 to 24.0]
Statistical Analysis 3: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Daily Activity Limitations - change to baseline to week 8; Test type: Superiority; p = 0.095, ANOVA; Least square mean difference = 16.4, 95% CI 2-sided [11.9 to 20.8]
Statistical Analysis 4: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 8; Test type: Superiority; p = 0.282, ANOVA; Least square mean difference = 14.5, 95% CI 2-sided [10.1 to 18.8]
Statistical Analysis 5: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Daily Activity Limitations - change from baseline to week 12; Test type: Superiority; p = 0.169, ANOVA; Least square mean difference = 15.0, 95% CI 2-sided [10.6 to 19.4]
Statistical Analysis 6: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 12; Test type: Superiority; p = 0.129, ANOVA; Least square mean difference = 15.4, 95% CI 2-sided [11.1 to 19.7]
Statistical Analysis 7: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Daily Activity Limitations - change from baseline to week 16; Test type: Superiority; p = 0.111, ANOVA; Least square mean difference = 14.0, 95% CI 2-sided [9.7 to 18.4]
Statistical Analysis 8: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 16; Test type: Superiority; p = 0.107, ANOVA; Least square mean difference = 14.0, 95% CI 2-sided [9.7 to 18.3]
Statistical Analysis 9: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Emotional Well-Being - change from baseline to week 4; Test type: Superiority; p = 0.827, ANOVA; Least square mean difference = 14.3, 95% CI 2-sided [9.7 to 18.9]
Statistical Analysis 10: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 4; Test type: Superiority; p = 0.688, ANOVA; Least square mean difference = 16.3, 95% CI 2-sided [11.8 to 20.8]
Statistical Analysis 11: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Emotional Well-Being - change from baseline to week 8; Test type: Superiority; p = 0.324, ANOVA; Least square mean difference = 15.7, 95% CI 2-sided [11.4 to 20.0]
Statistical Analysis 12: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 8; Test type: Superiority; p = 0.949, ANOVA; Least square mean difference = 12.9, 95% CI 2-sided [8.7 to 17.1]
Statistical Analysis 13: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Emotional Well-Being - change from baseline to week 12; Test type: Superiority; p = 0.927, ANOVA; Least square mean difference = 15.7, 95% CI 2-sided [11.4 to 20.1]
Statistical Analysis 14: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 12; Test type: Superiority; p = 0.776, ANOVA; Least square mean difference = 14.8, 95% CI 2-sided [10.8 to 18.8]
Statistical Analysis 15: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Emotional Well-Being - change from baseline to week 16; Test type: Superiority; p = 0.418, ANOVA; Least square mean difference = 15.7, 95% CI 2-sided [11.4 to 20.1]
Statistical Analysis 16: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 16; Test type: Superiority; p = 0.613, ANOVA; Least square mean difference = 14.8, 95% CI 2-sided [10.6 to 19.0]
Statistical Analysis 17: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Work Limitations - change from baseline to week 4; Test type: Superiority; p = 0.721, ANOVA; Least square mean difference = 15.8, 95% CI 2-sided [8.3 to 23.2]
Statistical Analysis 18: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Work Limitations - change from baseline to week 4; Test type: Superiority; p = 0.558, ANOVA; Least square mean difference = 20.6, 95% CI 2-sided [13.1 to 28.0]
Statistical Analysis 19: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Work Limitations - change from baseline to week 8; Test type: Superiority; p = 0.809, ANOVA; Least square mean difference = 18.4, 95% CI 2-sided [11.5 to 25.3]
Statistical Analysis 20: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Work Limitations - change from baseline to week 8; Test type: Superiority; p = 0.651, ANOVA; Least square mean difference = 19.4, 95% CI 2-sided [12.4 to 26.4]
Statistical Analysis 21: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Work Limitations - change from baseline to week 12; Test type: Superiority; p = 0.769, ANOVA; Least square mean difference = 16.4, 95% CI 2-sided [9.5 to 23.3]
Statistical Analysis 22: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Work Limitations - change from baseline to week 12; Test type: Superiority; p = 0.454, ANOVA; Least square mean difference = 21.3, 95% CI 2-sided [14.3 to 28.3]
Statistical Analysis 23: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Work Limitations - change from baseline to week 16; Test type: Superiority; p = 0.564, ANOVA; Least square mean difference = 18.3, 95% CI 2-sided [11.6 to 25.0]
Statistical Analysis 24: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Work Limitations - change from baseline to week 16; Test type: Superiority; p = 0.250, ANOVA; Least square mean difference = 21.0, 95% CI 2-sided [14.1 to 27.8]
Statistical Analysis 25: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment Satisfaction - change from baseline to week 4; Test type: Superiority; p = 0.853, ANOVA; Least square mean difference = 23.9, 95% CI 2-sided [15.6 to 32.2]
Statistical Analysis 26: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 4; Test type: Superiority; p = 0.393, ANOVA; Least square mean difference = 20.0, 95% CI 2-sided [11.9 to 28.0]
Statistical Analysis 27: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment Satisfaction - change from baseline to week 8; Test type: Superiority; p = 0.010, ANOVA; Least square mean difference = 27.9, 95% CI 2-sided [20.2 to 35.6]
Statistical Analysis 28: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 8; Test type: Superiority; p = 0.395, ANOVA; Least square mean difference = 18.3, 95% CI 2-sided [11.1 to 25.4]
Statistical Analysis 29: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment Satisfaction - change from baseline to week 12; Test type: Superiority; p = 0.068, ANOVA; Least square mean difference = 24.8, 95% CI 2-sided [17.1 to 32.4]
Statistical Analysis 30: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 12; Test type: Superiority; p = 0.400, ANOVA; Least square mean difference = 19.3, 95% CI 2-sided [12.2 to 26.4]
Statistical Analysis 31: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment Satisfaction - change from baseline to week 16; Test type: Superiority; p = 0.021, ANOVA; Least square mean difference = 25.5, 95% CI 2-sided [18.1 to 33.0]
Statistical Analysis 32: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 16; Test type: Superiority; p = 0.056, ANOVA; Least square mean difference = 23.1, 95% CI 2-sided [16.1 to 30.0]
Statistical Analysis 33: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment-Related Bother - change from baseline to week 4; Test type: Superiority; p = 0.981, ANOVA; Least square mean difference = 14.2, 95% CI 2-sided [7.6 to 20.7]
Statistical Analysis 34: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 4; Test type: Superiority; p = 0.525, ANOVA; Least square mean difference = 17.0, 95% CI 2-sided [11.1 to 22.9]
Statistical Analysis 35: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment-Related Bother - change from baseline to week 8; Test type: Superiority; p = 0.356, ANOVA; Least square mean difference = 9.5, 95% CI 2-sided [2.9 to 16.0]
Statistical Analysis 36: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 8; Test type: Superiority; p = 0.771, ANOVA; Least square mean difference = 6.5, 95% CI 2-sided [0.7 to 12.4]
Statistical Analysis 37: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment-Related Bother - change from baseline to week 12; Test type: Superiority; p = 0.926, ANOVA; Least square mean difference = 8.7, 95% CI 2-sided [2.0 to 15.5]
Statistical Analysis 38: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 12; Test type: Superiority; p = 0.778, ANOVA; Least square mean difference = 7.9, 95% CI 2-sided [1.9 to 13.9]
Statistical Analysis 39: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment-Related Bother - change from baseline to week 16; Test type: Superiority; p = 0.984, ANOVA; Least square mean difference = 10.0
Statistical Analysis 40: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 16; Test type: Superiority; p = 0.514, ANOVA; Least square mean difference = 7.4, 95% CI 2-sided [1.6 to 13.1]
Statistical Analysis 41: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Symptom Bother - change from baseline to week 4; Test type: Superiority; p = 0.985, ANOVA; Least square mean difference = -16.6, 95% CI 2-sided [-20.4 to -12.8]
Statistical Analysis 42: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 4; Test type: Superiority; p = 0.646, ANOVA; Least square mean difference = -17.8, 95% CI 2-sided [-21.5 to -14.0]
Statistical Analysis 43: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Symptom Bother - change from baseline to week 8; Test type: Superiority; p = 0.007, ANOVA; Least square mean difference = -20.7, 95% CI 2-sided [-24.5 to -16.9]
Statistical Analysis 44: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 8; Test type: Superiority; p = 0.305, ANOVA; Least square mean difference = -16.2, 95% CI 2-sided [-19.9 to -12.5]
Statistical Analysis 45: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Symptom Bother - change from baseline to week 12; Test type: Superiority; p = 0.015, ANOVA; Least square mean difference = -19.0, 95% CI 2-sided [-22.7 to -15.4]
Statistical Analysis 46: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 12; Test type: Superiority; p = 0.039, ANOVA; Least square mean difference = -18.0, 95% CI 2-sided [-21.5 to -14.4]
Statistical Analysis 47: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Test type: Superiority; p = 0.001, ANOVA; Least square mean difference = -19.7, 95% CI 2-sided [-23.3 to -16.0]
Statistical Analysis 48: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 16; Test type: Superiority; p = 0.002, ANOVA; Least square mean difference = -18.9, 95% CI 2-sided [-22.4 to -15.3]

16. Secondary Outcome: Change From Baseline in Quality of Life (Impact of Dry Eye on Everyday Life (IDEEL) Questionnaire vs Different Timepoints - Per Protocol Set
Description: as for outcome 15
Time Frame: At weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
score on a scale
  Daily activity limitations - Change from baseline to week 4 | 16.8 (21.20) | 19.7 (17.58) | 13.0 (20.63)
  Daily activity limitations - Change from baseline to week 8 | 17.1 (23.93) | 15.3 (16.85) | 11.5 (17.47)
  Daily activity limitations - Change from baseline to week 12 | 17.0 (20.30) | 16.5 (18.45) | 11.2 (17.64)
  Daily activity limitations - Change from baseline to week 16 | 13.9 (19.33) | 15.8 (19.74) | 9.4 (16.94)
  Emotional well-being - change from baseline to week 4 | 15.2 (21.73) | 17.3 (20.33) | 15.8 (20.60)
  Emotional well-being - change from baseline to week 8 | 16.9 (21.70) | 13.9 (18.34) | 13.2 (17.55)
  Emotional well-being - change from baseline to week 12 | 15.1 (18.58) | 16.4 (16.87) | 14.7 (18.14)
  Emotional well-being - change from baseline to week 16 | 16.8 (18.48) | 16.6 (18.59) | 14.2 (20.11)
  work limitations - change from baseline to week 4 | 16.0 (27.48) | 21.3 (24.83) | 18.4 (24.23)
  work limitations - change from baseline to week 8 | 17.4 (25.13) | 18.3 (19.43) | 17.9 (22.29)
  work limitations - change from baseline to week 12 | 15.0 (21.67) | 21.9 (21.82) | 18.6 (22.14)
  work limitations - change from baseline to week 16 | 15.4 (19.43) | 21.9 (20.93) | 16.7 (21.80)
  Treatment satisfaction/happiness - change from baseline to week 4 | 25.4 (31.05) | 19.6 (31.26) | 25.2 (33.81)
  Treatment satisfaction/happiness - change from baseline to week 8 | 30.1 (28.47) | 21.0 (27.85) | 13.9 (30.66)
  Treatment satisfaction/happiness - change from baseline to week 12 | 25.8 (31.16) | 21.6 (27.82) | 15.5 (26.81)
  Treatment satisfaction/happiness - change from baseline to week 16 | 26.0 (27.60) | 24.3 (28.26) | 13.2 (27.18)
  treatment-related bother - change from baseline to week 4 | 15.7 (22.66) | 15.3 (23.39) | 14.4 (27.71)
  treatment-related bother - change from baseline to week 8 | 11.6 (20.73) | 6.9 (25.46) | 4.6 (26.78)
  treatment-related bother - change from baseline to week 12 | 9.9 (22.83) | 10.0 (23.05) | 8.7 (28.26)
  treatment-related bother - change from baseline to week 16 | 11.4 (20.90) | 9.5 (21.62) | 9.8 (27.51)
  Dry eye symptom bother - change from baseline to week 4 | -17.3 (17.19) | -18.7 (16.64) | -17.2 (17.10)
  Dry eye symptom bother - change from baseline to week 8 | -21.5 (18.88) | -17.6 (15.40) | -13.9 (14.97)
  Dry eye symptom bother - change from baseline to week 12 | -19.6 (17.41) | -19.7 (17.16) | -13.2 (13.18)
  Dry eye symptom bother - change from baseline to week 16 | -20.6 (15.21) | -20.7 (17.66) | -11.3 (14.61)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Daily Activity Limitations - change from baseline to week 4; Test type: Superiority; p = 0.241, ANOVA; Least square mean difference = 16.8, 95% CI 2-sided [12.2 to 21.4]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 4; Test type: Superiority; p = 0.040, ANOVA; Least square mean difference = 19.7, 95% CI 2-sided [15.1 to 24.4]
Statistical Analysis 3: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Daily Activity Limitations - change from baseline to week 8; Test type: Superiority; p = 0.097, ANOVA; Least square mean difference = 16.8, 95% CI 2-sided [12.3 to 21.4]
Statistical Analysis 4: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 8; Test type: Superiority; p = 0.238, ANOVA; Least square mean difference = 15.3, 95% CI 2-sided [10.7 to 19.9]
Statistical Analysis 5: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Daily Activity Limitations - change from baseline to week 12; Test type: Superiority; p = 0.070, ANOVA; Least square mean difference = 16.5, 95% CI 2-sided [12.0 to 20.9]
Statistical Analysis 6: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 12; Test type: Superiority; p = 0.058, ANOVA; Least square mean difference = 16.7, 95% CI 2-sided [12.3 to 21.1]
Statistical Analysis 7: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Daily Activity Limitations - change from baseline to week 16; Test type: Superiority; p = 0.128, ANOVA; Least square mean difference = 13.7, 95% CI 2-sided [9.3 to 18.1]
Statistical Analysis 8: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Daily Activity Limitations - change from baseline to week 16; Test type: Superiority; p = 0.024, ANOVA; Least square mean difference = 16.0, 95% CI 2-sided [11.6 to 20.3]
Statistical Analysis 9: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Emotional Well-Being - change from baseline to week 4; Test type: Superiority; p = 0.865, ANOVA; Least square mean difference = 15.2, 95% CI 2-sided [10.4 to 20.1]
Statistical Analysis 10: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 4; Test type: Superiority; p = 0.662, ANOVA; Least square mean difference = 17.3, 95% CI 2-sided [12.4 to 22.2]
Statistical Analysis 11: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Emotional Well-Being - change from baseline to week 8; Test type: Superiority; p = 0.266, ANOVA; Least square mean difference = 16.7, 95% CI 2-sided [12.2 to 21.1]
Statistical Analysis 12: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 8; Test type: Superiority; p = 0.824, ANOVA; Least square mean difference = 13.9, 95% CI 2-sided [9.4 to 18.3]
Statistical Analysis 13: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Emotional Well-Being - change from baseline to week 12; Test type: Superiority; p = 0.883, ANOVA; Least square mean difference = 14.8, 95% CI 2-sided [10.6 to 19.0]
Statistical Analysis 14: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 12; Test type: Superiority; p = 0.516, ANOVA; Least square mean difference = 16.3, 95% CI 2-sided [12.1 to 20.4]
Statistical Analysis 15: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Emotional Well-Being - change from baseline to week 16; Test type: Superiority — Emotional Well-Being - change from baseline to week 16; p = 0.407, ANOVA; Least square mean difference = 16.5, 95% CI 2-sided [12.1 to 21.0]
Statistical Analysis 16: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Emotional Well-Being - change from baseline to week 16; Test type: Superiority; p = 0.422, ANOVA; Least square mean difference = 16.4, 95% CI 2-sided [12.0 to 20.9]
Statistical Analysis 17: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Work Limitations - change from baseline to week 4; Test type: Superiority; p = 0.615, ANOVA; Least square mean difference = 15.9, 95% CI 2-sided [8.1 to 23.8]
Statistical Analysis 18: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Work Limitations - change from baseline to week 4; Test type: Superiority; p = 0.626, ANOVA; Least square mean difference = 21.3, 95% CI 2-sided [13.3 to 29.2]
Statistical Analysis 19: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Work Limitations - change from baseline to week 8; Test type: Superiority; p = 0.968, ANOVA; Least square mean difference = 18.3, 95% CI 2-sided [11.1 to 25.6]
Statistical Analysis 20: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Test type: Superiority; p = 0.689, ANOVA; Least square mean difference = 20.1, 95% CI 2-sided [12.8 to 27.4]
Statistical Analysis 21: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Work Limitations - change from baseline to week 12; Test type: Superiority; p = 0.528, ANOVA; Least square mean difference = 15.6, 95% CI 2-sided [8.5 to 22.7]
Statistical Analysis 22: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Work Limitations - change from baseline to week 12; Test type: Superiority; p = 0.368, ANOVA; Least square mean difference = 23.0, 95% CI 2-sided [15.8 to 30.1]
Statistical Analysis 23: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Work Limitations - change from baseline to week 16; Test type: Superiority; p = 0.764, ANOVA; Least square mean difference = 17.7, 95% CI 2-sided [10.7 to 24.7]
Statistical Analysis 24: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Work Limitations - change from baseline to week 16; Test type: Superiority; p = 0.184, ANOVA; Least square mean difference = 22.6, 95% CI 2-sided [15.5 to 29.6]
Statistical Analysis 25: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment Satisfaction - change from baseline to week 4; Test type: Superiority; p = 0.909, ANOVA; Least square mean difference = 25.4, 95% CI 2-sided [16.5 to 34.2]
Statistical Analysis 26: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 4; Test type: Superiority; p = 0.428, ANOVA; Least square mean difference = 21.1, 95% CI 2-sided [12.2 to 30.0]
Statistical Analysis 27: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment Satisfaction - change from baseline to week 8; Test type: Superiority; p = 0.008, ANOVA; Least square mean difference = 29.8, 95% CI 2-sided [21.6 to 37.9]
Statistical Analysis 28: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 8; Test type: Superiority; p = 0.222, ANOVA; Least square mean difference = 21.3, 95% CI 2-sided [13.5 to 29.2]
Statistical Analysis 29: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Treatment Satisfaction - change from baseline to week 12; Test type: Superiority; p = 0.082, ANOVA; Least square mean difference = 25.3, 95% CI 2-sided [17.2 to 33.4]
Statistical Analysis 30: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 12; Test type: Superiority; p = 0.154, ANOVA; Least square mean difference = 23.3, 95% CI 2-sided [15.6 to 31.1]
Statistical Analysis 31: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment Satisfaction - change from baseline to week 16; Test type: Superiority; p = 0.030, ANOVA; Least square mean difference = 25.8, 95% CI 2-sided [18.0 to 33.6]
Statistical Analysis 32: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment Satisfaction - change from baseline to week 16; Test type: Superiority; p = 0.046, ANOVA; Least square mean difference = 24.6, 95% CI 2-sided [17.1 to 32.1]
Statistical Analysis 33: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; Treatment-Related Bother - change from baseline to week 4; Test type: Superiority; p = 0.861, ANOVA; Least square mean difference = 15.4, 95% CI 2-sided [8.6 to 22.2]
Statistical Analysis 34: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 4; Test type: Superiority; p = 0.865, ANOVA; Least square mean difference = 15.3, 95% CI 2-sided [9.0 to 21.7]
Statistical Analysis 35: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Treatment-Related Bother - change from baseline to week 8; Test type: Superiority; p = 0.278, ANOVA; Least square mean difference = 10.5, 95% CI 2-sided [3.6 to 17.3]
Statistical Analysis 36: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 8; Test type: Superiority; p = 0.689, ANOVA; Least square mean difference = 7.2, 95% CI 2-sided [0.9 to 13.5]
Statistical Analysis 37: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Treatment-Related Bother - change from baseline to week 12; Test type: Superiority; p = 0.993, ANOVA; Least square mean difference = 9.1, 95% CI 2-sided [2.1 to 16.2]
Statistical Analysis 38: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 12; Test type: Superiority; p = 0.989, ANOVA; Least square mean difference = 9.2, 95% CI 2-sided [2.8 to 15.7]
Statistical Analysis 39: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Treatment-Related Bother - change from baseline to week 16; Test type: Superiority; p = 0.976, ANOVA; Least square mean difference = 10.4, 95% CI 2-sided [3.7 to 17.0]
Statistical Analysis 40: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Treatment-Related Bother - change from baseline to week 16; Test type: Superiority; p = 0.778, ANOVA; Least square mean difference = 9.0, 95% CI 2-sided [2.9 to 15.1]
Statistical Analysis 41: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Symptom Bother - change from baseline to week 4; Test type: Superiority; p = 0.964, ANOVA; Least square mean difference = -17.3, 95% CI 2-sided [-21.2 to -13.3]
Statistical Analysis 42: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 4; Test type: Superiority; p = 0.581, ANOVA; Least square mean difference = -18.7, 95% CI 2-sided [-22.7 to -14.7]
Statistical Analysis 43: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Symptom Bother - change from baseline to week 8; Test type: Superiority; p = 0.006, ANOVA; Least square mean difference = -21.4, 95% CI 2-sided [-25.2 to -17.5]
Statistical Analysis 44: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 8; Test type: Superiority; p = 0.175, ANOVA; Least square mean difference = -17.6, 95% CI 2-sided [-21.4 to -13.7]
Statistical Analysis 45: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Symptom Bother - change from baseline to week 12; Test type: Superiority; p = 0.016, ANOVA; Least square mean difference = -19.4, 95% CI 2-sided [-23.1 to -15.6]
Statistical Analysis 46: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 12; Test type: Superiority; p = 0.010, ANOVA; Least square mean difference = -19.8, 95% CI 2-sided [-23.5 to -16.1]
Statistical Analysis 47: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; Symptom Bother - change from baseline to week 16; Test type: Superiority; p = 0.000, ANOVA; Least square mean difference = -20.5, 95% CI 2-sided [-24.3 to -16.8]
Statistical Analysis 48: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; Symptom Bother - change from baseline to week 16; Test type: Superiority; p = 0.000, ANOVA; Least square mean difference = -20.8, 95% CI 2-sided [-24.6 to -17.1]

17. Secondary Outcome: Patient Global Impression of Change (PGIC) - Full Analysis Set
Description: PGIC is a commonly used method of assessing clinically important change. With PGIC the qualitative assessment of meaningful change is determined by the patient on 7-items using a 0 (very much improved) to 10 (very much worse) scale.
Time Frame: At baseline and weeks 4, 8, 12 and 16
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
participants
  week 4 - Very Much Improved | 11 | 2 | 4
  week 4 - Much Improved | 18 | 15 | 20
  week 4 - Minimally improved | 18 | 21 | 20
  week 4 - no change | 24 | 38 | 38
  week 4 - minimally worse | 6 | 4 | 2
  week 4 - much worse | 1 | 1 | 0
  week 4 - very much worse | 0 | 0 | 0
  week 8 - Very much improved | 9 | 3 | 1
  week 8 - much improved | 23 | 11 | 16
  week 8 - minimally improved | 19 | 21 | 17
  week 8 - no change | 21 | 37 | 46
  week 8 - minimally worse | 1 | 4 | 2
  week 8 - much worse | 0 | 1 | 2
  week 8 - very much worse | 1 | 1 | 0
  week 12 - very much improved | 11 | 3 | 4
  week 12 - much improved | 16 | 10 | 12
  week 12 - minimally improved | 22 | 24 | 24
  week 12 - no change | 15 | 36 | 40
  week 12 - minimally worse | 5 | 1 | 0
  week 12 - much worse | 2 | 2 | 2
  week 12 - very much worse | 2 | 1 | 0
  week 16 - very much improved | 7 | 3 | 6
  week 16 - much improved | 24 | 19 | 16
  week 16 - minimally improved | 22 | 20 | 19
  week 16 - no change | 19 | 33 | 36
  week 16 - minimally worse | 2 | 2 | 5
  week 16 - much worse | 1 | 0 | 0
  week 16 - very much worse | 0 | 1 | 0
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; at week 4; Test type: Superiority; p = 0.302, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; at week 4; Test type: Superiority; p = 0.224, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; at week 8 (FUP); Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; at week 8 (FUP); Test type: Superiority; p = 0.885, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; At week 12 (FUP); Test type: Superiority; p = 0.035, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; At week 12 (FUP); Test type: Superiority; p = 0.698, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; At week 16 (FUP); Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; At week 16 (FUP); Test type: Superiority; p = 0.706, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Patient Global Impression of Change (PGIC) - Per Protocol Set
Description: as for outcome 17
Time Frame: At weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
participants
  week 4 - Very Much Improved | 10 | 2 | 4
  week 4 - Much Improved | 18 | 12 | 18
  week 4 - Minimally improved | 17 | 19 | 20
  week 4 - no change | 20 | 34 | 36
  week 4 - minimally worse | 6 | 4 | 2
  week 4 - much worse | 1 | 0 | 0
  week 4 - very much worse | 0 | 0 | 0
  week 8 - Very much improved | 9 | 3 | 1
  week 8 - much improved | 21 | 9 | 15
  week 8 - minimally improved | 18 | 21 | 17
  week 8 - no change | 20 | 34 | 43
  week 8 - minimally worse | 1 | 3 | 2
  week 8 - much worse | 0 | 1 | 2
  week 8 - very much worse | 0 | 0 | 0
  week 12 - very much improved | 11 | 3 | 4
  week 12 - much improved | 13 | 9 | 11
  week 12 - minimally improved | 21 | 23 | 23
  week 12 - no change | 15 | 33 | 38
  week 12 - minimally worse | 5 | 1 | 0
  week 12 - much worse | 2 | 1 | 2
  week 12 - very much worse | 1 | 0 | 0
  week 16 - very much improved | 7 | 3 | 6
  week 16 - much improved | 22 | 18 | 15
  week 16 - minimally improved | 19 | 17 | 18
  week 16 - no change | 19 | 30 | 34
  week 16 - minimally worse | 2 | 2 | 5
  week 16 - much worse | 0 | 0 | 0
  week 16 - very much worse | 0 | 0 | 0
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; at week 4; Test type: Superiority; p = 0.210, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; at weeek 4; Test type: Superiority; p = 0.260, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; At week 8 (FUP); Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; at week 8 (FUP); Test type: Superiority; p = 0.734, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; at week 12 (FUP); Test type: Superiority; p = 0.050, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; at week 12 (FUP); Test type: Superiority; p = 0.985, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; at week 16 (FUP); Test type: Superiority; p = 0.018, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; at week 16 (FUP); Test type: Superiority; p = 0.580, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Change From Baseline in EQ-5D-3L Questionnaire to Different Timepoints - Full Analysis Set
Description: EQ-5D is a standardised measure of health status. - The EQ-5D 3 level version (EQ-5D-3L) consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS) which are summed up.
  The EQ-5D-3L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. This scale ranges from 5 (best case) to 15 (worst case).
  Each dimension has 3 levels: no problems, some problems, extreme problems (labelled 1-3). The respondent must indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  - The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This is a quantitative measure of health outcome, judged by each respondent.
  Both for total and partial scores, the higher the score, the worse is the outcome.
Time Frame: At weeks 4, 8, 12 and 16
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 81 | 82 | 84
score on a scale
  week 4 | 1.2 (9.91) | 3.8 (10.28) | 2.8 (8.86)
  week 8 | 2.7 (10.41) | 2.4 (8.92) | 2.1 (8.86)
  week 12 | 3.0 (10.10) | 3.0 (7.8) | 3.0 (8.59)
  week 16 | 3.0 (13.04) | 4.8 (11.92) | 2.0 (11.71)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; statistical analysis at week 4; Test type: Superiority; p = 0.282, ANOVA; Least square mean difference = 1.2, 95% CI 2-sided [-1.0 to 3.3]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 4; Test type: Superiority; p = 0.497, ANOVA; Least square mean difference = 3.9, 95% CI 2-sided [1.7 to 6.0]
Statistical Analysis 3: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; statistical analysis at week 8; Test type: Superiority; p = 0.734, ANOVA; Least square mean difference = 2.6, 95% CI 2-sided [0.5 to 4.8]
Statistical Analysis 4: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 8; Test type: Superiority; p = 0.963, ANOVA; Least square mean difference = 2.2, 95% CI 2-sided [0.1 to 4.3]
Statistical Analysis 5: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; statistical analysis at week 12; Test type: Superiority; p = 0.854, ANOVA; Least square mean difference = 2.7, 95% CI 2-sided [0.7 to 4.8]
Statistical Analysis 6: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 12; Test type: Superiority; p = 0.881, ANOVA; Least square mean difference = 2.8, 95% CI 2-sided [0.8 to 4.8]
Statistical Analysis 7: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; statistical analysis at week 16; Test type: Superiority; p = 0.632, ANOVA; Least square mean difference = 3.0, 95% CI 2-sided [0.3 to 5.7]
Statistical Analysis 8: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 16; Test type: Superiority; p = 0.220, ANOVA; Least square mean difference = 4.4, 95% CI 2-sided [1.7 to 7.0]

20. Secondary Outcome: Change From Baseline in EQ-5D-3L Questionnaire to Different Timepoints - Per Protocol Set
Description: as for outcome 19
Time Frame: Aat baseline and weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rhNGF 20 μg/ml TID | rhNGF 20 μg/ml BID + Vehicle OD | Vehicle TID
Number analyzed (Participants) | 72 | 71 | 80
score on a scale
  week 4 | 1.2 (9.98) | 3.6 (8.12) | 2.8 (8.99)
  week 8 | 2.7 (10.67) | 2.3 (9.02) | 2.2 (8.79)
  week 12 | 3.6 (9.77) | 3.4 (5.00) | 3.0 (8.71)
  week 16 | 3.3 (13.24) | 4.7 (8.84) | 1.9 (11.90)
Statistical Analysis 1: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; statistical analysis at week 4; Test type: Superiority; p = 0.296, ANOVA; Least square mean difference = 1.2, 95% CI 2-sided [-0.9 to 3.3]
Statistical Analysis 2: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 4; Test type: Superiority; p = 0.570, ANOVA; Least square mean difference = 3.6, 95% CI 2-sided [1.5 to 5.7]
Statistical Analysis 3: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; statistical analysis at week 8; Test type: Superiority; p = 0.754, ANOVA; Least square mean difference = 2.7, 95% CI 2-sided [0.5 to 4.9]
Statistical Analysis 4: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 8; Test type: Superiority; p = 0.972, ANOVA; Least square mean difference = 2.3, 95% CI 2-sided [0.0 to 4.5]
Statistical Analysis 5: Comparison: rhNGF 20 μg/ml TID vs rhNGF 20 μg/ml BID + Vehicle OD; statistical analysis at week 12; Test type: Superiority; p = 0.793, ANOVA; Least square mean difference = 3.4, 95% CI 2-sided [1.4 to 5.3]
Statistical Analysis 6: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 12; Test type: Superiority; p = 0.766, ANOVA; Least square mean difference = 3.4, 95% CI 2-sided [1.5 to 5.3]
Statistical Analysis 7: Comparison: rhNGF 20 μg/ml TID vs Vehicle TID; statistical analysis at week 16; Test type: Superiority; p = 0.458, ANOVA; Least square mean difference = 3.3, 95% CI 2-sided [0.6 to 6.0]
Statistical Analysis 8: Comparison: rhNGF 20 μg/ml BID + Vehicle OD vs Vehicle TID; statistical analysis at week 16; Test type: Superiority; p = 0.147, ANOVA; Least square mean difference = 4.6, 95% CI 2-sided [2.0 to 7.3]

ADVERSE EVENTS:
Time Frame: From Screening day to week 16
Description: More specifically, adverse events are assessed at Screening day, Visit 1 Day 1), Visit 2 (Day 14), Visit 3 (Day 28), Visit 4 (Day 56), Visit 5 (Day 84), Visit 6 (Day 112).
Groups:
- rhNGF 20 μg/ml TID - Treatment Period; rhNGF 20 μg/ml TID - Follow-up Period: One drop of rhNGF 20 μg/ml will be instilled in both eyes three times daily (every 6-8 hours)
  rhNGF 20 μg/ml: one drop of rhNGF 20 μg/ml will be instilled in both eyes three times daily (every 6-8 hours)
- rhNGF 20 μg/ml BID + Vehicle OD - Treatment Period; rhNGF 20 μg/ml BID + Vehicle OD - Follow-up Period: One drop of rhNGF 20 μg/ml will be instilled in both eyes two times daily (BID) plus one drop (40 μL) of vehicle will be instilled in both eyes once daily (OD) (every 6-8 hours)
  rhNGF 20 μg/ml + vehicle: one drop of rhNGF 20 μg/ml will be instilled in both eyes two times daily plus one drop (40 μL) of vehicle will be instilled in both eyes once daily (every 6-8 hours).
  rhNGF will be instilled in the morning and in the evening while the vehicle will be instilled in the afternoon.
- Vehicle TID - Treatment Period; Vehicle TID - Follow up Period: Vehicle eye one drop will be instilled in both eyes three times daily (every 6-8 hours)
  Vehicle: one drop of vehicle will be instilled in both eyes three times daily (every 6-8 hours)
Arm/Group | rhNGF 20 μg/ml TID - Treatment Period | rhNGF 20 μg/ml BID + Vehicle OD - Treatment Period | Vehicle TID - Treatment Period | rhNGF 20 μg/ml TID - Follow-up Period | rhNGF 20 μg/ml BID + Vehicle OD - Follow-up Period | Vehicle TID - Follow up Period
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/84 | 0/88 | 0/85 | 0/84 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/84 | 0/88 | 1/85 | 0/84 | 1/88
Other Adverse Events (participants affected / at risk) | 65/85 | 60/84 | 26/88 | 19/85 | 19/84 | 18/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20 μg/ml TID - Treatment Period (N=85) | rhNGF 20 μg/ml BID + Vehicle OD - Treatment Period (N=84) | Vehicle TID - Treatment Period (N=88) | rhNGF 20 μg/ml TID - Follow-up Period (N=85) | rhNGF 20 μg/ml BID + Vehicle OD - Follow-up Period (N=84) | Vehicle TID - Follow up Period (N=88)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20 μg/ml TID - Treatment Period (N=85) | rhNGF 20 μg/ml BID + Vehicle OD - Treatment Period (N=84) | Vehicle TID - Treatment Period (N=88) | rhNGF 20 μg/ml TID - Follow-up Period (N=85) | rhNGF 20 μg/ml BID + Vehicle OD - Follow-up Period (N=84) | Vehicle TID - Follow up Period (N=88)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Conjunctival Disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (2) | 3 (3) | 5 (6) | 2 (2) | 0 (0) | 1 (1)
Erythema Of Eyelid (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Eye Allergy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye Discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 2 (2) | 5 (14) | 5 (6) | 1 (1) | 2 (5) | 4 (4)
Eye Pain (Eye disorders) | 54 (68) | 42 (73) | 4 (5) | 1 (1) | 1 (1) | 1 (1)
Eye Pruritus (Eye disorders) | 2 (4) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Eye Swelling (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid Disorder (Eye disorders) | 1 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid Irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eyelid Oedema (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid Pain (Eye disorders) | 3 (6) | 9 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign Body Sensation In Eyes (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meibomian Gland Dysfunction (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ocular Discomfort (Eye disorders) | 6 (9) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 2 (2) | 3 (4) | 3 (4) | 2 (2) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Posterior Capsule Opacification (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Refraction Disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling Of Eyelid (Eye disorders) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 3 (3) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 2 (2)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation Site Irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation Site Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory Tract (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial Injury Of Eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 5 (5) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine With Aura (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder Prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03982368/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03982368/SAP_001.pdf